CLINICAL TRIAL: NCT03994653
Title: Cancer Loyalty Card Study: a Retrospective Observational Case-Control Study
Brief Title: Cancer Loyalty Card Study
Acronym: CLOCS
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Cancer Research UK (Other); Imperial College Healthcare NHS Trust (Other); Sandwell & West Birmingham Hospitals NHS Trust (Other); University College London Hospitals (Other); County Durham and Darlington NHS Foundation Trust (Other Government); Walsall Healthcare NHS Trust (Other); Surrey and Sussex Healthcare NHS Trust (Other); Airedale NHS Foundation Trust (Other); Abertawe Bro Morgannwg University Health Board (Other); Gateshead Health NHS Foundation Trust (Other); Norfolk and Norwich University Hospitals NHS Foundation Trust (Other); The Leeds Teaching Hospitals NHS Trust (Other); NHS Lothian (Other Government); East Lancashire Hospitals NHS Trust (Other); University Hospitals Bristol and Weston NHS Foundation Trust (Other); Royal Surrey County Hospital NHS Foundation Trust (Other); Royal Marsden NHS Foundation Trust (Other); Velindre NHS Trust (Other Government); Cardiff and Vale University Health Board (Other Government); South Tees Hospitals NHS Foundation Trust (Other); West Hertfordshire Hospitals NHS Trust (Other); The Christie NHS Foundation Trust (Other); Manchester University NHS Foundation Trust (Other Government); NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Other Study IDs: 19IC5156
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Results first posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Ovarian Neoplasms
Keywords: Ovarian cancer; Cancer of the ovary; Observational study; Case-control study; Cancer Loyalty Card Study; CLOCS
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Participants diagnosed with ovarian cancer
  Interventions: Other: Risk Factor Questionnaire; Other: Clinical Questionnaire
- Controls: Participants without ovarian cancer
  Interventions: Other: Risk Factor Questionnaire

INTERVENTIONS:
Other: Risk Factor Questionnaire — For cases, the study recruiter at the Trust will present this in the clinic. Controls will complete this online or at home when volunteering to participate. The participant questionnaire will be completed by the participant.
  Other Names: Participant Questionnaire
Other: Clinical Questionnaire — For cases, the study recruiter at the trust will complete this form together with the participant. Controls will not complete this form.
  Groups: Cases

SUMMARY:
Approximately 7,400 new cases of ovarian cancer are diagnosed each year in the United Kingdom (UK), and with over 4,000 women dying from the disease each year it is a particularly lethal form of cancer. The symptoms for ovarian cancer are not well known and vague, and most women are diagnosed at a late stage when the cancer has already spread around the abdominal cavity with poor prognosis. Novel methods are needed to improve earlier detection and thereby improve survival from this disease.

The Cancer Loyalty Card Study (CLOCS) proposes to use loyalty card data from two participating high street retailers to investigate purchase behaviour as an opportunity for cancer symptom surveillance. The investigators aim to conduct a case-control study of ovarian cancer patients matched with women without ovarian cancer and to explore public preferences for how to communicate potential outcomes of the commercial and health data linkages back to individuals.

Eligible participants will be women in the UK who own at least one loyalty card with the participating high street retailers. Of these women, those who have been diagnosed with ovarian cancer are eligible to participate in the study as cases, while women who have not been diagnosed with ovarian cancer are eligible to participate as controls.

Upon choosing to participate, all participants will be asked to complete a short questionnaire about well-established ovarian cancer risk factors and common symptoms either in the clinic (cases) or online/from a packet in the mail(controls). This information will be used in risk assessment for ovarian cancer of participants, which will be used at the analysis stage.

DETAILED DESCRIPTION:
Purpose and Design

The Cancer Loyalty Card Study (CLOCS) is addressing whether or not data already collected by high street retailers can detect significant changes in purchase behaviours of ovarian cancer patients prior to their diagnosis. The investigators aim to conduct a case-control study of ovarian cancer patients matched with women who do not have ovarian cancer. The study aims to recruit at least 500 recently diagnosed ovarian cancer patients and at least 500 healthy women as controls and collate up to 7 years of prior purchase data.

This is a database only study.

Recruitment

Loyalty card holders will be invited to join the study by email and post from the high street retailers and can choose to sign up via the CLOCS website or via post by returning the consent form to the study team through the mail. There will also be a press release about the study inviting loyalty card holders to visit the CLOCS website for more information and join the study. Women, 18 years or older, who have a loyalty card at the participating high street retailers are eligible to join. Women with ovarian cancer and who own at least one of the participating high street retailer's loyalty cards will be recruited in a clinic by a member of their healthcare team where the study is open. Any woman considering joining the study can contact the research team using the contact details on the information sheet.

Consent

Ovarian cancer patients will be given the information sheet and consent form in the clinic by a member of their healthcare team. They can take as much time as they need to read through the information sheet. If they choose to participate, they can complete the consent form whenever is convenient for them and return it to the CLOCS team in the free post envelope provided to them in the clinic.

Women without ovarian cancer will be presented with the information sheet and consent form in an email or letter in the mail from their high street retailer if they hold a loyalty card with them and return them to the CLOCS team in a free post envelope. They can also find the information sheet and consent form on the CLOCS website and consent online.

Methods

Consenting participants will complete a brief questionnaire about ovarian cancer risk factors, which will also be returned to the CLOCS team through the mail or on the website (healthy volunteers only). Participants with ovarian cancer will also have a clinical form for a member of their clinical team to complete in the clinic. This will be sent to the CLOCS team along with their consent and risk factor questionnaire in the free post envelope. Two ovarian cancer patients have reviewed all questionnaires and CLOCS documents and expressed their approval. Women without ovarian cancer from the general UK population have also reviewed the risk factor questionnaire and expressed their approval saying the questionnaire is 'easy to understand' and 'straightforward'.

If participants consent to be re-contacted by the CLOCS team for future studies or for loyalty card detail clarification,they will provide either a contact email or phone number. There is no further action needed from participants once they complete their consent form and questionnaire (and clarify loyalty card details if necessary)

ELIGIBILITY:
Inclusion Criteria:

* Women, at least 18 years old, recently diagnosed with ovarian cancer (preferably recruited just after diagnosis and during treatment period,but are still eligible if diagnosed up to 2 years prior, at the latest) who hold at least one participating high street retailer loyalty card are eligible to join the CLOCS as cases.

Women, at least 18 years old, who have not been diagnosed with ovarian cancer and hold at least one participating high street retailer loyalty card are eligible to join the CLOCS as controls.

Exclusion Criteria:

* Women under the age of 18 years and, since this is a study about ovarian cancer,men will not be eligible to join this study. Women who do not own loyalty cards with the participating high street retailers are not eligible to join this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Ovarian cancer is a female only cancer.
Study Population: All participants will be females in the UK who are at least 18 years old and who own at least one of the participating high street retailer loyalty cards. Participants who have been diagnosed with ovarian cancer are considered cases. Participants who do not have ovarian cancer are considered controls.
Sampling Method: Non-Probability Sample
Enrollment: 963 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Flanagan, PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Only aggregated and anonymised survey data will be shared with other researchers after publication. No sensitive individual level data will be shared.

REFERENCES:
- [Background] Flanagan JM, Skrobanski H, Shi X, Hirst Y. Self-Care Behaviors of Ovarian Cancer Patients Before Their Diagnosis: Proof-of-Concept Study. JMIR Cancer. 2019 Jan 17;5(1):e10447. doi: 10.2196/10447. PMID 30664464
- [Result] Brewer HR, Chadeau-Hyam M, Johnson E, Sundar S, Flanagan J, Hirst Y. Cancer Loyalty Card Study (CLOCS): feasibility outcomes for an observational case-control study focusing on the patient interval in ovarian cancer. BMJ Open. 2023 Jun 14;13(6):e066022. doi: 10.1136/bmjopen-2022-066022. PMID 37316316
- [Derived] Brewer HR, Hirst Y, Chadeau-Hyam M, Johnson E, Sundar S, Flanagan JM. Association Between Purchase of Over-the-Counter Medications and Ovarian Cancer Diagnosis in the Cancer Loyalty Card Study (CLOCS): Observational Case-Control Study. JMIR Public Health Surveill. 2023 Jan 26;9:e41762. doi: 10.2196/41762. PMID 36701184
- [Derived] Brewer HR, Hirst Y, Sundar S, Chadeau-Hyam M, Flanagan JM. Cancer Loyalty Card Study (CLOCS): protocol for an observational case-control study focusing on the patient interval in ovarian cancer diagnosis. BMJ Open. 2020 Sep 8;10(9):e037459. doi: 10.1136/bmjopen-2020-037459. PMID 32900761

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The target enrolment for this study was 1000. However, the study enrolled 963 participants (306 cases and 657 controls).
  609 participants remained after confirming first part of eligibility (182 cases and 427 controls).
  273 participants remained after confirming second part of eligibility (153 cases and 120 controls)
Period: Overall Study
Arm/Group | Cases | Controls
Started | 306 | 657
Completed | 153 (153 cases met all eligibility for the study) | 120 (120 controls met all eligibility for the study)
Not Completed | 153 | 537

BASELINE CHARACTERISTICS:
Population: From the 306 cases, 183 cases returned their questionnaires and one was excluded.
  From 657 controls, 230 were excluded for not meeting the inclusion criteria, other reasons (duplicate test submissions) and withdrawl.
  Participant numbers as per Table 1
Groups:
- Total: Total of all reporting groups
Arm/Group | Cases | Controls | Total
Number analyzed (Participants) | 182 | 427 | 609
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 98 | 368 | 466
  >=65 years | 84 | 59 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (10.9) | 51.6 (13.7) | 55.5 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182 | 427 | 609
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 181 | 411 | 592
  Unknown or Not Reported | 1 | 16 | 17
Region of Enrollment [Number; unit: participants]
  United Kingdom | 182 | 427 | 609

OUTCOME MEASURES:

1. Primary Outcome: Purchase Behaviours (Purchase of Items)
Description: The primary outcome of the CLOCS will be to define the time by which the cases and controls are statistically significantly (p=0.05) different in their purchase behaviours leading up to ovarian cancer diagnosis. A higher purchase amount of relevant items (pain and indigestion medications) in cases compared to controls associated with cancer.
Time Frame: 24 months
Population: All participants for whom loyalty card data was received (cases and controls)
Measure: Mean (Standard Deviation); unit: number of items purchased
Arm/Group | Cases | Controls
Number analyzed (Participants) | 153 | 120
number of items purchased
  6 months (0-6) | 3.2 (8.4) | 2.0 (3.0)
  12 months (0-12) | 5.9 (13.6) | 4.3 (6.3)
  24 months (0-24) | 11.4 (25.0) | 8.5 (11.4)
Statistical Analysis 1: Comparison: Cases vs Controls; Fishers exact test, conducted at each month prior to diagnosis comparing total purchases of relevant products (pain and indigestion medication) compared with all purchases in both cases and controls. Power calculation: we used a power calculation assuming the Fisher Exact Test to calculate the minimum group size to detect a difference in purchase proportions that we hypothesised with 80% statistical power; Test type: Superiority; p < 0.001, Fisher Exact; Odds Ratio (OR) = 2.91, 95% CI 2-sided [2.07 to 4.12]

2. Secondary Outcome: Alert About Cancer Symptoms Assessed by Purchase Behaviour
Description: The secondary outcome of the CLOCS will be defining a purchase threshold as an "alert" about cancer symptoms in individuals
Time Frame: 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: There were no adverse events to collect as there was no intervention.
Description: No adverse events were collected as this was an observational study with no interventions. Therefore, all events are 0 as this was not applicable to our study. The study did not collect information on any adverse events related or not related to the disease or any medical treatment administered as part of their standard of care.
Groups:
- Cases; Controls: no adverse event data was collected as this was an observational study.
Arm/Group | Cases | Controls
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-06): https://cdn.clinicaltrials.gov/large-docs/53/NCT03994653/Prot_SAP_000.pdf